CLINICAL TRIAL: NCT04825730
Title: Long-Term Extension Study of Investigator Initiated Trial to Evaluate Cartilage Regeneration by Arthroscopy in Patients With K-L Grade III Knee Osteoarthritis After 『JOINTSTEM』 Administration
Brief Title: Follow-up Study for Participants of Jointstem Investigator Initiated Trial by Arthroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BS-JS-IIT1-FU
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Degenerative Arthritis; Knee Arthritis
Keywords: Stem cell; Adipose tissue derived mesenchymal stem cell; Osteoarthritis; degenerative arthritis; long term; Biostar; Rbio
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long Term Follow-up after Jointstem Transplantation (Experimental)
  Interventions: Drug: JOINTSTEM

INTERVENTIONS:
Drug: JOINTSTEM — JOINTSTEM is an OA treatment that uses autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissues and is incubated without additional genetic modification or mechanical and chemical modification through differentiation, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.
  Other Names: autologous adipose-derived mesenchymal stem cells

SUMMARY:
This clinical trial is conducted to assess the long-term safety of "jointstem" in patients with degenerative knee arthritis who participated in the previous BS-JS-IIT1 investigator initiated trial.

DETAILED DESCRIPTION:
JOINTSTEM is injectables for an OA treatment that uses autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissues and is cultured without additional genetic modification, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.

This clinical trial is planned to follow-up the long-term safety of "jointstem" in patients with degenerative knee arthritis who participated in the previous BS-JS-IIT1 investigator initiated trial.

Subjects who participate in the BS-JS-IIT1 study and agree to this extension test in writing will be assessed for safety by conducting laboratory tests, vital signs, physical examinations and adverse events every 12 months after Visit 1.

However, after unblinding of the BS-JS-IIT1 investigator initiated trial, subjects in the control group (placebo administration) will terminate the follow-up of this extended clinical trial and conduct routine treatment for degenerative knee arthritis at the discretion of the researcher. Appropriate measures and follow-up observations shall be implemented for abnormal reactions occurred during this extended test period until they are terminated (such as the loss of the relevant adverse event or inability to conduct follow-up investigations).

ELIGIBILITY:
Inclusion Criteria:

* Participants of Jointstem IIT by arthroscopy (BS-JS-IIT1)
* Participants who signed informed consent document of this study

Exclusion Criteria:

* No applicable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 60 Month
  Incidence of adverse events from baseline to 60 months

SECONDARY OUTCOMES:
Adverse Events (Special Attention Target) | 60 months
  Incidence of adverse events(special attention target: malicious tumor, autoimmune disease) from baseline to 60 months

IPD SHARING:
Plan to Share IPD: No